CLINICAL TRIAL: NCT07359664
Title: Optical Coherence Tomography Angiography (OCTA) for the Assessment of Retinal Capillary Density in Patients With Cardiovascular Disease and a Healthy Control Group
Brief Title: OCTA in Cardiovascular Disease and Healthy Controls
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: German Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OCTA_CVD
Record Dates: First submitted 2025-12-09; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Patients With Cardiovascular Disease; Healthy Participants
Keywords: arterial hypertension; type 2 diabetes mellitus; chronic kidney disease; heart failure
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Heart Failure

STUDY DESIGN:
Intervention Model Description: Assessment of OCTA and SLDF in all patients/healthy individuals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment of retinal vessels (Other): OCTA and SLDF based assessment of retinal vasculature
  Interventions: Diagnostic Test: Retinal vascular assessment using OCTA and SLDF

INTERVENTIONS:
Diagnostic Test: Retinal vascular assessment using OCTA and SLDF — Assessment of retinal capillary density using OCTA and SLDF

SUMMARY:
This prospective clinical study will involve the non-invasive assessment of retinal vessels using OCTA (Cirrus OCT 6000 AngioPlex) and scanning laser Doppler flowmetry (SLDF) in patients with cardiovascular disease and healthy individuals. The study will be conducted at the Clinical Research Centre (CRC), Department of Nephrology and Hypertension at the University of Erlangen-Nuremberg.

DETAILED DESCRIPTION:
Each patient (32 patients) and healthy individual (32 healthy individuals) undergoes one study visit. After providing informed consent, each patient and healthy individual receives an assessment of their retinal vessels using OCTA and SLDF. In the sub-study of 10 patients with cardiovascular disease, the reliability of the OCTA measurements will be determined. Each patient will receive three study visits (with an OCTA and SLDF assessment on each occasion) on three different days.

ELIGIBILITY:
Inclusion Criteria for patients with cardiovascular disease:

* cardiovascular disease defined as one or more of the following: arterial hypertension, type 2 diabetes mellitus, chronic kidney disease, heart failure

Inclusion Criteria for healthy individuals:

* BMI 18-29.9 kg/m2
* Non-smoker
* Good general health, as determined by study personnel based on assessments of previous visits, including anamnesis, vital signs, physical examination and clinical laboratory parameters.

Exclusion criteria for patients with cardiovascular disease:

* Active ophthalmological (retinal) disease resulting in impaired visual assessment of retinal vessels (e.g. glaucoma, cataracts, retinal oedema).

Exclusion criteria for healthy individuals:

* Active ophthalmological (retinal) disease with reduced visual assessment of retinal vessels (e.g. glaucoma, cataracts, retinal oedema).
* clinically relevant deviation in physical examination, vital signs, or laboratory parameters (based on the physician's clinical judgement).
* a clinically relevant history of cardiovascular disease or any other previously known cardiovascular disease
* History of clinically relevant neurological, gastrointestinal, renal, hepatic, psychological, pulmonary, metabolic, endocrine or other diseases
* office blood pressure above or equal to 140/90 mmHg
* Office heart rate outside of the following range: 50-99 bpm
* regular intake of any medication for the treatment of cardiovascular diseases (e.g. antihypertensive or antidiabetic medication) within one month before study inclusion
* alcohol or drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of reliability of OCTA based assessment of retinal capillary density in patients with CV disease | test-retest-reliability between 3 study visits (between each visit needs to be a time gap of at least 24 hours, all visits will be performed within two weeks)
  Assessment of test-retest-reliability between 3 study visits for OCTA based assessment of retinal capillary density in patients with CV disease

SECONDARY OUTCOMES:
comparison of OCTA based retinal capillary density between CV diseased patients and healthy controls | one study visit in each group, baseline values at day 1 are compared
  comparison of OCTA based retinal capillary density between CV diseased patients and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Bosch, MD, Principal Investigator — Clinical Research Center, Department of Nephrology and Hypertension, Universityhospital Erlangen
Locations (1):
- University of Erlangen Nuremberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No